CLINICAL TRIAL: NCT00977652
Title: Short Term Efficacy of Percutaneous Tibial Nerve Stimulation for the Treatment of Fecal Incontinence:Randomized Controlled Study
Brief Title: Percutaneous Tibial Nerve Stimulation for the Treatment of Fecal Incontinence
Acronym: TENSIA
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University Hospital, Rouen (Other)
Collaborators: Ministry of Health, France (Other Government)
Responsible Party: Principal Investigator, Anne Marie LEROI, Head of the department, University Hospital, Rouen
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2008/070/HP; CPP-2008/032; RCB-2008-A01227-48
Record Dates: First submitted 2009-09-15; First posted 2009-09-16 (Estimated); Last update posted 2011-08-23 (Estimated); Status verified 2011-08

CONDITIONS: Fecal Incontinence
Keywords: fecal incontinence
MeSH Terms: conditions — Fecal Incontinence

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Active stimulation (Active Comparator): Percutaneous posterior tibial nerve stimulation
  Interventions: Procedure: active stimulation
- sham stimulation (Sham Comparator): Inefficient percutaneous posterior tibial nerve stimulation
  Interventions: Procedure: sham stimulation

INTERVENTIONS:
Procedure: active stimulation — percutaneous posterior tibial nerve stimulation with following parameters: frequency: 14hz; impulse duration: 210usec;intensity:sensibility threshold during 3 months
  Arms: Active stimulation
Procedure: sham stimulation — Same location with the same device than active stimulation but amplitude of stimulation = 0
  Arms: sham stimulation

SUMMARY:
Fecal incontinence is a major public health issue since 10% of the French population aged 45 has to deal with it. Different treatments exist and have already been evaluated, like the sacral nerve stimulation (SNS) which has proved to be efficient in 75 to 100% of the anal incontinence patients without significant sphincteric lesions or rectal prolapse. However, the treatment is expensive and can have side effects. Moreover, about 20 to 30% of the patients can develop a resistance to the SNS only a few months following the definite implantation. Yet the development of the posterior tibial nerve stimulation (PNTS) offers a new perspective. It consists in stimulating the same metameric area as the sacral nerves. It is regularly used for the treatment of urinary incontinence caused by overactive bladder. It is a non-invasive technique, causing but a few side effects. A preliminary study showed that 7 in 10 incontinent patients saw an improvement when treated with PTNS.

Purpose:

The aim of this study is to analyse and evaluate the PTNS technique in the short term as a treatment of anal incontinence. It is done through the means of a multi-centric prospective randomized study.

Patients:

Will be included: all patients followed for anal incontinence (either with liquid or solid stools) having at least one accident a month for 3months, and who are not diagnosed with colorectal lesions and who are without anal or rectal significant anatomic anomalies, without rectal prolapse, and who have failed to respond to medical treatment (such as medicine or perineal reeducation). The main criterium to analyze the efficiency will be the number of fecal incontinence episodes on a bowel diary. The investigators aim to incorporate 144 patients, that is 72 in each group. 12 centers will take part in this study, that will last 2 years and 3 months. They are the centers of: Bordeaux, Clermont-Ferrand, Grenoble, Lyon, Marseille, Nancy, Nantes, Paris, Diaconesses-Croix,Paris Rothschild, Rennes, Rouen, and Toulouse.

Method:

The PTNS consists in setting two electrodes on the posterial tibial nerve pathway. The electrodes are connected to an external stimulator. After having drawn lots, patients will be treated for 3months either with effective stimulation (frequency: 14hz; impulse duration: 210usec;intensity:sensibility threshold), or with shame stimulation (intensity: 0mAmp). There will be two daily sessions of stimulation (effective, or shame), 20 min each. A pre-treatment assessment will be established, composed of a stool diary, a Cleveland Clinic score, a Fecal Incontinence Quality of Life scale and an anorectal manomety, that will all be repeated by the end of the treatment.

Expected Results:

The investigators hope to prove the short term efficacy of the PTNS on anal incontinence patients.

ELIGIBILITY:
Inclusion Criteria:

* fecal incontinence, refractory to medical treatment,for more than 3 months,with at least one episode of anal incontinence and/or urgency per month
* patient with no knowledge of cutaneous stimulation
* patients with NHS

Exclusion Criteria:

* older than 18 years old
* pregnancy
* implanted stimulator
* cutaneous lesion
* cutaneous anesthesia
* patients without oral contraception
* Guardianship and curatorship
* fecal incontinence secondary to anorectal malformation, surgical sequelae, significative sphincteric lesion leading to repair at a first time, rectal prolapse, active neurological disease
* patient already treated by sacral nerve stimulation or stimulated graciloplasty, artificial bowel sphincter, radiofrequency

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 144 (Estimated)
Dates: Start 2009-10; Primary Completion 2011-06 (Actual); Study Completion 2011-06 (Actual)

PRIMARY OUTCOMES:
fecal incontinence episode per week | three months

SECONDARY OUTCOMES:
cleveland clinic score FIQL score analogic visual scale urinary score and anorectal manometry | 3 months

CONTACTS AND LOCATIONS:
Locations (1):
- Leroi, Rouen, France